CLINICAL TRIAL: NCT03848208
Title: A Phase I, Double-blind, Randomized, Placebo-controlled, Single Dose-escalation Study to Evaluate the Tolerability and Safety of Cytisine in Adult Smokers
Brief Title: A Single Dose-escalation Study of Cytisine in Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-CYT-08; 2018-003344-22 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Cohort 1: Cytisine 6.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 1: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 2: Cytisine 9.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 2: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 3: Cytisine 12.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 3: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 4: Cytisine 15.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 4: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 5: Cytisine 18.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 5: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 6: Cytisine 21.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 6: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 7: Cytisine 24.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 7: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 8: Cytisine 27.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 8: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo
- Cohort 9: Cytisine 30.0 mg (Experimental): Cytisine will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: cytisine
- Cohort 9: Placebo (Placebo Comparator): Placebo will be administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cytisine — cytisine film-coated oral tablet
  Other Names: Tabex; cytisinicline
  Arms: Cohort 1: Cytisine 6.0 mg; Cohort 2: Cytisine 9.0 mg; Cohort 3: Cytisine 12.0 mg; Cohort 4: Cytisine 15.0 mg; Cohort 5: Cytisine 18.0 mg; Cohort 6: Cytisine 21.0 mg; Cohort 7: Cytisine 24.0 mg; Cohort 8: Cytisine 27.0 mg; Cohort 9: Cytisine 30.0 mg
Drug: placebo — matching placebo oral tablet
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo; Cohort 6: Placebo; Cohort 7: Placebo; Cohort 8: Placebo; Cohort 9: Placebo

SUMMARY:
The objectives of this study are:

1. To assess the tolerability and safety of cytisine as a single oral dose.
2. To define the Cmax levels associated to the occurrence of dose-limiting adverse events.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following criteria to be eligible for inclusion into the study:

1. Free written informed consent prior to any procedure required by the study.
2. Male or female subjects, age ≥18 years, at the time of signing the informed consent.
3. Current daily cigarette smokers (averaging at least 10 cigarettes per day in the past 30 days).
4. Expired air carbon monoxide (CO) ≥10 ppm.
5. Able to swallow multiple tablets at one time.
6. Able to fully understand, comply with all study requirements.

Exclusion Criteria:

Subjects meeting ANY of the following exclusion criteria will NOT be eligible for inclusion into the study at screening.

1. Known hypersensitivity to cytisine or any of the excipients.
2. Known severe hypersensitivity to any other drug.
3. Positive urinary drugs of abuse screen, determined within 28 days before cytisine/placebo dosing.
4. Positive ethanol breath test.
5. Clinically significant abnormal serum chemistry, hematology, coagulation or urinalysis values within 28 days of randomization (i.e. requiring treatment or monitoring).
6. Clinically significant abnormalities in 12-lead echocardiogram (ECG) determined after minimum of 5 minutes in supine position within 28 days of randomization (i.e. requiring treatment or further assessment).
7. Body Mass Index (BMI) classification for being underweight (<18.5 kg/m2) or having ≥Class 2 obesity (≥35 kg/m2).
8. History of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident, cardiac arrhythmia, or hospitalization for congestive heart failure.
9. Blood pressure ≥160/100 mmHg, measured on the dominant arm, after at least 3 minutes in supine position.
10. Creatinine clearance (CrCl) <80 mL/min (estimated with the Cockroft-Gault equation).
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 x the upper limit of normal (ULN).
12. Any inability to comply with study restrictions (See Section 9)
13. Any inability or difficulty in fasting.
14. Difficulty in donating blood on either arm.
15. If woman of childbearing potential, positive result in serum beta-human chorionic gonadotropin (hCG) pregnancy test.
16. Women who are breast-feeding.
17. Subjects who do not agree to use acceptable methods of birth control during the study (See Section 9.4).
18. Participation in a clinical study with an investigational drug within the previous 2 months.
19. Participation in more than 2 clinical trials within the previous 12 months.
20. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

    Subjects meeting ANY of the following exclusion criteria will NOT be eligible for inclusion into the study at admission to each cohort.
21. Any recent disease or condition or treatment that, according to the Investigator, would put the subject at undue risk due to study participation.
22. Positive urinary drugs of abuse screen.
23. Positive ethanol breath test.
24. If female of childbearing potential, positive result in urine beta-hCG pregnancy test.
25. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Hospital da Prelada
Locations (1):
- BlueClinical, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a single center in Portugal.
Pre-assignment Details: Participants were randomly assigned to receive a single oral dose of cytisine or placebo in a 3:1 ratio (6 cytisine:2 placebo) for each dose cohort. Seventy-four (74) participants were randomized; 2 were withdrawn from the study by physician decision before dosing (1 due to high blood pressure and 1 due to noncompliance with protocol restrictions).
Groups:
- Placebo: Placebo to match Cytisine 6-30 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 6 mg: Cytisine 6 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 9 mg: Cytisine 9 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 12 mg: Cytisine 12 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 15 mg: Cytisine 15 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 18 mg: Cytisine 18 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 21 mg: Cytisine 21 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 24 mg: Cytisine 24 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 27 mg: Cytisine 27 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
- Cytisine 30 mg: Cytisine 30 mg administered in the morning, orally, with 240 mL of water, after fasting overnight for at least 10 hours.
Period: Overall Study
Arm/Group | Placebo | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg
Started (randomized and treated) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.5) | 44.5 (12.1) | 35.7 (8.2) | 35.3 (11.1) | 34.7 (7.5) | 37.8 (12.9) | 30.3 (8.1) | 30.0 (5.5) | 30.3 (4.6) | 29.7 (8.9) | 33.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 2 | 2 | 3 | 2 | 2 | 2 | 1 | 0 | 28
  Male | 8 | 2 | 4 | 4 | 3 | 4 | 4 | 4 | 5 | 6 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 71
  Multiple Races | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Study Discontinuation
Description: An adverse event (AE) is defined as any untoward medical occurrence that does not necessarily have to have a causal relationship with the treatment. A serious AE is any untoward medical occurrence or effect, that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; or is an important medical event which requires medical intervention to prevent one of the above. Treatment emergent events are those that occurred after the first dose of study drug.
Time Frame: From first dose of study drug through Day 6
Population: Safety Set: all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Any TEAE | 5 | 2 | 1 | 4 | 3 | 2 | 1 | 2 | 2 | 4
  Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1: Pre-dose (within 30 minutes prior to dosing), 15, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, and 3 hours (+/-2 minutes) post-dose
Population: Pharmacokinetic Analysis Set: all participants who received a dose of cytisine and had evaluable pharmacokinetic data.
Measure: Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 71.05 [56.07 to 86.03] | 93.62 [79.44 to 107.79] | 94.27 [74.87 to 113.66] | 126.45 [100.82 to 152.07] | 134.94 [107.00 to 162.88] | 150.08 [114.12 to 186.04] | 171.44 [149.31 to 193.57] | 151.05 [122.01 to 180.08] | 166.65 [120.95 to 212.34]

3. Primary Outcome: Pharmacokinetics: Time to Occurrence of Cmax (Tmax)
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set: all participants who received a dose of cytisine and had evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.83 [0.50 to 2.00] | 1.38 [0.83 to 2.50] | 1.88 [1.25 to 2.50] | 1.88 [0.50 to 2.50] | 2.00 [1.50 to 3.00] | 1.89 [1.25 to 3.00] | 2.50 [0.83 to 3.00] | 2.75 [1.75 to 3.00] | 2.50 [1.00 to 3.00]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Day 6
Arm/Group | Placebo | Cytisine 6 mg | Cytisine 9 mg | Cytisine 12 mg | Cytisine 15 mg | Cytisine 18 mg | Cytisine 21 mg | Cytisine 24 mg | Cytisine 27 mg | Cytisine 30 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/18 | 2/6 | 1/6 | 4/6 | 3/6 | 2/6 | 1/6 | 2/6 | 2/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Cytisine 6 mg (N=6) | Cytisine 9 mg (N=6) | Cytisine 12 mg (N=6) | Cytisine 15 mg (N=6) | Cytisine 18 mg (N=6) | Cytisine 21 mg (N=6) | Cytisine 24 mg (N=6) | Cytisine 27 mg (N=6) | Cytisine 30 mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03848208/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03848208/SAP_001.pdf